CLINICAL TRIAL: NCT05688345
Title: Comparison of Recovery Profiles of Propofol, Dexmedetomidine, and Remimazolam for Monitored Anesthetic Care in Patients Undergoing Upper Limb Surgery Under Brachial Plexus Block : a Randomized Controlled Trial
Brief Title: Comparison of Recovery Profiles Among Propofol, Remimazolam, and Dexmedetomidine After Intraoperative Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hajung Kim, clinical assistant professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-1591
Record Dates: First submitted 2022-12-30; First posted 2023-01-18 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Remimazolam; Propofol; Dexmedetomidine; Orthopedic Procedures; Sedatives; Brachial Plexus Block
MeSH Terms: interventions — remimazolam; Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remimazolam (Active Comparator): Maintenance doses of remimazolam is administered for sedation
  Interventions: Drug: Remimazolam
- Propofol (Active Comparator): Propofol is administered for sedation through target-controlled infusion
  Interventions: Drug: Propofol
- Dexmedetomidine (Active Comparator): Loading and maintenance doses of dexmedetomidine are administered for sedation
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Remimazolam — The patient receives continuous infusion of remimazolam at a rate of 0.3-1.0 mg/kg/hr.
  Arms: Remimazolam
Drug: Propofol — Patients are administered propofol at an effective site concentration of 1.0-2.5 mcg/ml through target-controlled infusion.
  Arms: Propofol
Drug: Dexmedetomidine — The patient is administered a dose of dexmedetomidine at 1 mcg/kg for 10 minutes, followed by continuous infusion at a rate of 0.2-1.0 mcg/kg/hr.
  Arms: Dexmedetomidine

SUMMARY:
A total of 120 patients (American Society of Anesthesiologist Physical Status 1-3) who signed a consent form among patients aged 19-80 years who are scheduled to undergo brachial plexus block and upper extremity surgery under monitored anesthetic care at our hospital were enrolled.

Recruited patients are divided into three groups through computer-generated randomization by using the patient identification number assigned during patient recruitment. (40 people in each group) Standard monitoring is performed when the patient arrives at the operating room. Patients receive oxygen at 5-6 L/min using a simple facial mask, and receive a brachial plexus block under ultrasound guidance. After confirming the success of brachial plexus block, administration of propofol, remimazolam, or dexmedetomidine is started according to the assigned group. Assess the patient's level of consciousness through the MOAA/S (modified observer's assessment of alertness/sedation scale) scale. The drug injection ends when the skin suture is started after the main procedure. The time from the end of injection of each drug until MOAA/S becomes 5 points is measured. After the patient is transferred to the recovery room, the Aldrete score is assessed.

The recovery profile, perioperative hemodynamic change, desaturation event, block duration, patient movement during surgery, patient satisfaction, and surgeon's satisfaction were investigated and analyzed for comparison.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS 1-3
* Patients scheduled for upper extremity surgery under brachial plexus block and monitored anesthetic care

Exclusion Criteria:

* Patients who refuse to participate in this study
* Patients with poorly controlled hypertension, hyperthyroidism, or moderate to severe heart disease
* Patients with severe hepatic or renal disease
* Patients who are chronically using antidepressants, anticonvulsants, or psychoactive drugs
* Patients who abuse drugs or alcohol
* Patients with severe sleep apnea
* Patients with cognitive impairment who have severe difficulties in communication
* Patients with allergy to propofol, dexmedetomidine, or remimazolam
* Patients judged to be inappropriate for this study

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2023-08-13 (Actual)

PRIMARY OUTCOMES:
Recovery profile | up to 1 hour after post-anesthesia case unit entry
  Time taken for MOAA/S score to reach 5 (MOAA/S: Modified Observer's Alertness/Sedation scale) Awake (5) - Unresponsive (0)

SECONDARY OUTCOMES:
Length of stay in post-anesthesia care unit | up to 3 hours after post-anesthesia case unit entry
  Length of stay from entering PACU to leaving
Intraoperative hypotension | up to 1hour from the initiation of sedative administration
  mean blood pressure less than 60mmHg
Occurrence of desaturation during surgery | From the start of sedative injection to the end of surgery or assessed up to 3 hours
  Oxygen saturation less than 92%
Duration of nerve block | From end of surgery until 24 hours after end of surgery
patient satisfaction | From end of surgery until 24 hours after end of surgery
  7 point Likert scale
Surgeon's satisfaction | From end of surgery until 24 hours after end of surgery
  7 point Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim HJ, Kim YJ, Lee J, Jeong D, Shin YH, Ro YJ, Kim H, Koh WU. Comparison of the recovery profiles of propofol, dexmedetomidine, and remimazolam for intraoperative sedation in patients undergoing upper limb surgery under brachial plexus blockade: a randomized controlled trial. Can J Anaesth. 2025 Jul;72(7):1090-1100. doi: 10.1007/s12630-025-02987-3. Epub 2025 Jun 13. PMID 40514628